CLINICAL TRIAL: NCT02366676
Title: Efficacy of Combined Intravesical Therapy With Hyaluronic Acid and Chondroitin Sulphate in the Treatment of Recurrent Cystitis Refractory to Escherichia Coli Extract: a Multicenter, Prospective Study
Brief Title: Efficacy of IARULIL® in the Treatment of Recurrent Cystitis Refractory to Escherichia Coli Extract
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-07-170
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Recurrent Cystitis
Keywords: Recurrent cystitis; hyaluronic acid; chondroitin sulphate
MeSH Terms: conditions — Cystitis | interventions — Hyaluronic Acid; Chondroitin; chondroitin sulfate, sodium hyaluronate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment group (Experimental): -Intervention: combined intravesical therapy with hyaluronic acid and chondroitin sulphate(IALURIL®) ( 1st month: once a week, 2nd~5th month:once a month)
  Interventions: Drug: hyaluronic acid and chondroitin sulphate

INTERVENTIONS:
Drug: hyaluronic acid and chondroitin sulphate — IALURIL Intravesical instillation with cystoscope ( 1st month: once a week, 2nd~5th month:once a month)
  Other Names: IALURIL®

SUMMARY:
The purpose of this study is to evaluate the efficacy of Combined Intravesical Therapy With Hyaluronic Acid and Chondroitin Sulphate in the Treatment of Recurrent Cystitis Refractory to Escherichia Coli Extract

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of combined intravesical therapy with hyaluronic acid and chondroitin sulphate(IARULIL®) in the treatment of recurrent cystitis refractory to oral Escherichia Coli extract(Uro-Vaxom®) and the change of urinary tract infection symptoms after intravesical instillation treatment with IARULIL®.

ELIGIBILITY:
Inclusion Criteria:

1. female patients aged between 20 and 80 years
2. Patients diagnosed with recurrent cystitis and treated with Escherichia Coli Extract
3. Patients with Refractory to Escherichia Coli Extract treatment

Exclusion Criteria:

1. child-bearing potential, pregnant or nursing women.
2. Residual urine volume >100ml
3. genitourinary tuberculosis or cancer / anatomical abnomality of genitourinary tract / neurologic abnormality of low urinary tract.
4. history of treatment for acute cystitis within 2weeks.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
The number of recurrence for recurrent cystitis | 12 months

SECONDARY OUTCOMES:
Time interval of cystitis | 12months
The score change of UTI symptom Assessment questionnaire(UTISA) | 12months
Global Respone assessment(GRA) score assessment | 12 month after treatment
safety evaluation Safety evaluation | 12 month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea